CLINICAL TRIAL: NCT01039116
Title: Taking Action Together: Development, Implementation and Evaluation of Community-Based Programs That Aims to Reduce Risk of Type 2 Diabetes in High BMI African American Children.
Brief Title: Taking Action Together- A Diabetes Prevention Program
Acronym: TAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sharon E Fleming, Principal Investigator, University of California at Berkeley
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: USDA 2004-35215-14250
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2007-03

CONDITIONS: Type 2 Diabetes
Keywords: obesity; nutrition; type 2 diabetes; community-based.
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Ultrasonic Waves

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Level of intervention intensity (Experimental): High Intensity: Behavioral Experimental:Participating children were invited to attend a 2 week summer day camp at the beginning of each intervention year, and to attend a weekly, 2 hr interactive session for children. Activities provided hand-on experiences preparing and tasting healthy food alternatives, engaging in a range of physical activities and self-esteem boosting via activities that promoted communication and positive behavioral development.
  Active Comparator: Low-intensity Participants were provided with educational materials 4 times yearly.
  Interventions: Behavioral: High Intensity; Behavioral: Low Intensity

INTERVENTIONS:
Behavioral: High Intensity — High-intensity intervention, Experimental. Participating children were invited to attend a 2 week summer day camp at the beginning of each intervention year, and to attend a weekly, 2 hr interactive session for children. Activities provided hand-on experiences preparing and tasting healthy food alternatives, engaging in a range of physical activities and self-esteem boosting via activities that promoted communication and positive behavioral development.
Behavioral: Low Intensity — Low-intensity intervention, Active comparator. Participants were provided with educational materials 4 times yearly.

SUMMARY:
The purpose of this study was to determine whether once-weekly exposure to a program that fostered self-esteem building, and improvements in nutrition and physical activity behaviors would reduce risk of type 2 diabetes in overweight, inner-city, African American children when compared to a control group.

DETAILED DESCRIPTION:
In the United States and, indeed, worldwide the prevalence of overweight and obesity has increased at an unprecedented rate. Concomitant with this demographic change are increases in diseases including type 2 diabetes, cardiovascular disease and some cancers that are associated with body fatness. Strategies to reduce body weight have been largely unsuccessful, making it unlikely that our population will be made healthy simply by recommending that overweight people reduce their body fatness. There is evidence, however, that the impact of body fat on human health can be significantly attenuated by potentially achievable strategies. Such strategies require adequate intakes of essential nutrients, regular physical activity and strong self-esteem. The goal of the project is to reduce the risk of type 2 diabetes mellitus (T2DM) in overweight 9- to 10-year-old African American children through a multi-component community-based program. The specific objectives are to (1).Implement a randomly controlled 2-phase intervention involving a 2-week summer camp, and weekly & monthly reinforcement sessions over 2 years, that include nutrition education, physical activity promotion, and self-esteem and self-efficacy building and (2) Test effectiveness of the program after 1 and 2 years of intervention on insulin sensitivity, the primary outcome, and on secondary outcomes including body fatness, dietary intakes, physical activity, and self-esteem. Identifying an effective, community-based program that could reduce risk of type 2 diabetes in high-risk children would promote health, reduce disease and reduce health-care costs in the future.

ELIGIBILITY:
Inclusion Criteria:

* Child age of 9-10 yr old at baseline
* Child BMI at least 85th percentile when matched for age and gender
* Able and willing to participate in normal daily activities
* Living in inner-city regions of Oakland CA

Exclusion Criteria:

* Fasting blood glucose of 120 mg/dl or higher
* Diagnosis of diabetes or other central metabolic disease
* Taking medications that interfere with or treat main study outcomes

Ages: 9 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2005-03; Primary Completion 2008-08 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
1 Year change in insulin resistance via HOMA-IR | Change during first year
  Baseline HOMA-IR minus Year 1 HOMA-IR
2 year change in insulin resistance via HOMA-IR | Change during 2 years
  Baseline HOMA-IR minus Year 2 HOMA-IR

SECONDARY OUTCOMES:
Change in dietary intakes of energy, fat, carbohydrate and selected essential nutrients. Change in minutes/day spend in moderate- and high-intensity physical activity. Improvement or stabilization of self-esteem. | 3years

CONTACTS AND LOCATIONS:
Overall Officials: Sharon E Fleming, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- YMCA of the East Bay, Oakland, CA 94612, Oakland, California, United States

REFERENCES:
- [Result] Raman A, Fitch MD, Hudes ML, Lustig RH, Murray CB, Ikeda JP, Fleming SE. Baseline correlates of insulin resistance in inner city high-BMI African-American children. Obesity (Silver Spring). 2008 Sep;16(9):2039-45. doi: 10.1038/oby.2008.329. PMID 19186328
- [Result] Raman A, Lustig RH, Fitch M, Fleming SE. Accuracy of self-assessed Tanner staging against hormonal assessment of sexual maturation in overweight African-American children. J Pediatr Endocrinol Metab. 2009 Jul;22(7):609-22. doi: 10.1515/jpem.2009.22.7.609. PMID 19774842
- [Result] Sharma S, Roberts LS, Hudes ML, Lustig RH, Fleming SE. Macronutrient intakes and cardio metabolic risk factors in high BMI African American children. Nutr Metab (Lond). 2009 Oct 13;6:41. doi: 10.1186/1743-7075-6-41. PMID 19825190
- [Result] Raman A, Sharma S, Fitch MD, Fleming SE. Anthropometric correlates of lipoprotein profile and blood pressure in high BMI African American children. Acta Paediatr. 2010 Jun;99(6):912-9. doi: 10.1111/j.1651-2227.2009.01639.x. Epub 2010 Jan 7. PMID 20064141
- [Result] Susan Stone,Aarthi Raman, Sharon Fleming.Behavioral characteristics among obese/overweight inner-city African American Children: A secondary analysis of participants in a community-based Type 2 diabetes risk reduction program. Children and Youth Services Review 32 (2010)833-839. doi:10.1016/j.childyouth.2010.02.002
- [Result] Sharma S, Roberts LS, Lustig RH, Fleming SE. Carbohydrate intake and cardiometabolic risk factors in high BMI African American children. Nutr Metab (Lond). 2010 Feb 9;7(1):10. doi: 10.1186/1743-7075-7-10. PMID 20181134
- [Result] Raman A, Ritchie LD, Lustig RH, Fitch MD, Hudes ML, Fleming SE. Insulin resistance is improved in overweight African American boys but not in girls following a one-year multidisciplinary community intervention program. J Pediatr Endocrinol Metab. 2010 Jan-Feb;23(1-2):109-20. doi: 10.1515/jpem.2010.23.1-2.109. PMID 20432814
- [Result] Ritchie LD, Sharma S, Ikeda JP, Mitchell RA, Raman A, Green BS, Hudes ML, Fleming SE. Taking Action Together: a YMCA-based protocol to prevent type-2 diabetes in high-BMI inner-city African American children. Trials. 2010 May 21;11:60. doi: 10.1186/1745-6215-11-60. PMID 20492667
- [Result] Sharma S, Lustig RH, Fleming SE. Identifying metabolic syndrome in African American children using fasting HOMA-IR in place of glucose. Prev Chronic Dis. 2011 May;8(3):A64. Epub 2011 Apr 15. PMID 21477504
- [Result] Fyfe M, Raman A, Sharma S, Hudes ML, Fleming SE. Insulin resistance and self-perceived scholastic competence in inner-city, overweight and obese, African American children. Physiol Behav. 2011 Jan 10;102(1):36-41. doi: 10.1016/j.physbeh.2010.09.015. Epub 2010 Sep 29. PMID 20887741
- [Derived] Sharma S, Fleming SE. One-year change in energy and macronutrient intakes of overweight and obese inner-city African American children: effect of community-based Taking Action Together type 2 diabetes prevention program. Eat Behav. 2012 Aug;13(3):271-4. doi: 10.1016/j.eatbeh.2012.03.003. Epub 2012 Mar 29. PMID 22664410
- See also: Taking Action Together: Overview and Curriculum — http://cwh.berkeley.edu/sites/default/files/primary_pdfs/Taking_Action_Together_Overview_Resources_ALL_0.pdf